CLINICAL TRIAL: NCT05339958
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of a Nutraceutical Supplement With Standardized Botanicals in Males With Self-Perceived Thinning Hair
Brief Title: Nutraceutical Supplement With Standardized Botanicals in Males With Thinning Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceutical Wellness Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NW-MS-03
Record Dates: First submitted 2022-04-04; First posted 2022-04-21 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Hair Thinning
Keywords: Nutraceutical; Supplement
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: This is a 6-month, multi-center, randomized, double-blind, placebo-controlled study in adult male subjects with self-perceived hair thinning. Subjects will be randomly assigned to either Nutrafol® Men hair growth supplement or placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutraceutical Dietary Supplement Capsule (Experimental): The nutraceutical capsules are comprised of standardized, natural, medical-grade ingredients. Subject will be instructed to take four (4) capsules by mouth once daily with a substantial meal.
  Interventions: Dietary Supplement: Nutrafol® Men Hair Growth Nutraceutical
- Placebo Capsule (Placebo Comparator): The placebo capsules contain no active ingredients. Subject will be instructed to take four (4) capsules by mouth once daily with a substantial meal.
  Interventions: Other: Placebo Supplement

INTERVENTIONS:
Dietary Supplement: Nutrafol® Men Hair Growth Nutraceutical — Nutrafol® Men contains patented Synergen Complex® is a blend of proprietary formulation of botanicals with potent anti-inflammatory, anti-stress adaptogenic, antioxidant and DHT-inhibiting properties - combined to synergistically combat the multiple underlying factors that compromise hair growth and health. These ingredients include Sensoril Ashwagandha, BCM-95 BioCurcumin, USPlus Saw Palmetto, EVNolMax 20% Tocotrienol/Tocopherol complex, Bioperine (piperine), Cynatine HNS (solubilized keratin), and Capsimax (capsaicin).
  Arms: Nutraceutical Dietary Supplement Capsule
Other: Placebo Supplement — The placebo capsules contain no active ingredients.
  Arms: Placebo Capsule

SUMMARY:
The objective of this study is to assess the effectiveness and safety of a novel dietary supplement containing botanical ingredients for hair thinning in men over the course of six months of continuous daily usage.

DETAILED DESCRIPTION:
Hair thinning is a common condition affecting both men and women that is more recently understood to be the result of multiple causes. Although it is generally a benign condition, hair thinning can have a significant, detrimental impact on self-esteem, psychosocial functioning and the overall quality of life of affected individuals. It can also represent a substantial financial burden on individuals seeking treatment.

The objective of this randomized, double-blind, placebo-controlled study is to assess the effectiveness and safety of a novel dietary supplement containing botanical ingredients for hair thinning over the course of six months of continuous daily usage. The study supplement is scientifically formulated to specifically target the multiple underlying causes of hair thinning. In addition to the necessary vitamins, minerals, and proteins to support the nutritional needs of hair, it also contains clinically tested, standardized pharmaceutical-grade botanicals (substances obtained from plants) that target hormones, stress and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Males between 21-55 years of age with self-perceived thinning
* Voluntarily sign and date an informed consent agreement and photo release form approved by the Institutional Review Board
* Clinically confirmed to have hair thinning or loss by the investigator or qualified sub-investigator via physical exam, including only subjects with male pattern hair loss with frontal and/or vertex patterns II, IIA, III, IIIv and IV using the Norwood classification of patterned hair loss in males.
* General good health, as determined by the Investigator or qualified sub-investigator
* Willing and able to attend all study visits and comply with the test product daily instructions.
* Willing to maintain the same hair style and same color for the duration of the study.
* Willing to use a mild non-medicated shampoo and conditioner for the duration of the study (medicated shampoo and conditioner refer to any prescription shampoo or conditioner as well as any over-the counter medicated shampoo or conditioner, such as those for treatment of dandruff or promoting hair growth).
* Willing and able to cooperate with the requirements of the study.
* Able to complete and understand the various rating instruments.

Exclusion Criteria:

* Individuals who have experienced serious complications due to COVID-19 previously or during the study as determined by the investigator.
* Clinical diagnosis of hair loss disorder such as alopecia areata, or scarring forms of alopecia.
* Subjects with male pattern hair loss with frontal and/or vertex patterns I, IIIA, IVA, V, VA, VI, VII using the Norwood classification of patterned hair loss in males.
* Scalp hair loss on the treatment area, due to disease, injury, or medical therapy
* Current skin disease (e.g., psoriasis, atopic dermatitis, skin cancer, eczema, sun damage, seborrheic dermatitis), cuts and or abrasions on the scalp or condition (e.g., sunburn, tattoos) on the treatment area that, in the opinion of the Investigator or qualified sub-investigator, might put the subject at risk or interfere with the study conduct or evaluations.
* History of surgical correction of hair loss on the scalp (i.e. hair transplant).
* Use of any products or devices purported to promote scalp hair growth (e.g., finasteride or minoxidil) within the 6 months prior to the Baseline Visit.
* Use of anti-androgenic therapies (e.g., spironolactone, flutamide, cyproterone acetate, progesterone, and bicalutamide) within 3 months prior to the Baseline Visit.
* History of burning, flaking, itching, and stinging of the scalp.
* History of malignancy (except cutaneous squamous cell carcinoma and basal cell carcinoma) or currently undergoing chemotherapy or radiation treatments.
* A known history of autoimmune thyroid disease, any other thyroid disorder/abnormality or other autoimmune disorders that in the opinion of the Investigator or qualified sub-investigator may interfere with the study treatment.
* A known history of unstable or chronic depression or bipolar disease or any other condition that may impact the subject's participation in the opinion of the investigator or qualified sub-investigator.
* A known allergy to any of the ingredients in the investigational product.
* Utilization of low-level lasers for hair growth in the last three months.
* Any condition that the Investigator thinks may put the subject at risk or interfere with their participation in the study.
* Known history or recent blood work indicating iron deficiency, bleeding disorders or platelet dysfunction syndrome as well as subjects receiving anticoagulant therapy or smokers with usage >20 cigarettes/day.
* Use of any medications or medicated shampoos that are known to potentially cause hair loss or affect hair growth, as determined by the Investigator or qualified sub-investigator.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 112 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Change in terminal hair counts | Day 180
  Changes in terminal hair counts as measured by photorichogram

SECONDARY OUTCOMES:
Proportion of subjects with ≥5% hair growth | Day 180
Change in total, terminal and vellus and hair count | Day 180
  Changes in all hair counts as measured by photorichogram
Change in mean hair width and mean inter-follicular distance | Day 180
  Changes in hair measurements as measured by photorichogram
Change in terminal to vellus ratio | Day 180
  Changes in hair ratio as measured by photorichogram
Change in mean number of hairs per follicular unit | Day 180
  Changes in hair density as measured by photorichogram
Hair Shedding | Day 180
  Change in Numbers of Hairs Shedded in Hair Pull Test
Subject Assessments | Day 180
  Subject self assessments of improvement in hair thickness and quality, quality of life, stress, and perception of the study product using questionnaires
Blinded Investigator Assessment | Day 180
  Changes in Investigator Hair Quality Global Improvement Scale & Investigator Hair Growth Global Improvement Scale assessed by physician using standardized 2-D photographs compared to baseline.
Compiled side effects | Day 180
  All side effects, including all expected or unexpected side effects, categorized by severity (Mild, moderate, severe) and relatedness to the study product or participation

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ablon Skin Institute and Research Center, Manhattan Beach, California
  - Therapeutic Clinical Research, San Diego, California

IPD SHARING:
Plan to Share IPD: No